CLINICAL TRIAL: NCT01976299
Title: AVERT™ Clinical Trial
Brief Title: AVERT™ Clinical Trial for Contrast Media Volume Reduction and Incidence of CIN
Acronym: AVERT™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osprey Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TP-6364
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Contrast Induced Nephropathy (CIN)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment (Experimental): Standard of Care with the AVERT system
  Interventions: Device: AVERT
- Standard of Care (No Intervention)

INTERVENTIONS:
Device: AVERT
  Arms: Active Treatment

SUMMARY:
The Osprey Medical AVERT System is indicated to reduce contrast media (CM) exposure to the kidneys during percutaneous coronary procedures thereby reducing the risk of contrast induced nephropathy (CIN).

DETAILED DESCRIPTION:
The purpose of this trial is to assess the AVERT System device, which is designed to limit the volume of CM (Contrast Media) utilized, during a staged therapeutic coronary PCI (Percutaneous Coronary Intervention) or a coronary diagnostic procedure that is anticipated to become a PCI (i.e. ad hoc PCI) for the reduction of CIN (Contrast Induced Nephropathy).

ELIGIBILITY:
Inclusion Criteria:

* The subject is a candidate for a therapeutic percutaneous coronary intervention (PCI) procedure.
* The subject has documented chronic kidney disease (CKD)

Exclusion Criteria:

* Subject is in acute renal failure
* Assessment of ventricular function that cannot be accomplished without the use of the CM.
* Subject has acute STEMI within 72 hours prior to planned PCI procedure, or is currently having an acute STEMI.
* Subject is unable to undergo peri-procedural hydration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Mehran, MD, FACC, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (39):
- United States (37):
  - UCSD Medical Center, La Jolla, California
  - Long Beach CA VA Hospital, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Stanford Hospital and Clinics, Stanford, California
  - Harbor UCLA Medical Center, Torrance, California
  - The Heart & Vascular Institute of Florida, Clearwater, Florida
  - University of FL College of Medicine - Jacksonville, Jacksonville, Florida
  - St. Vincent's Ambulatory Care (dba St. Vincent's Cardiology), Jacksonville, Florida
  - Tallahassee Research Institute, Inc., Tallahassee, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - St. Joseph's Hospital (Emory), Atlanta, Georgia
  - Coliseum Medical Center, Macon, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Jewish Hospital, Louisville, Kentucky
  - Norton Cardiovascular Associates, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Minneapolis Heart Institute Foundation / Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic Hospital, St. Mary's Campus, Rochester, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Saint Luke's Hospital, Kansas City, Missouri
  - Gateway Cardiovascular Research Center, Inc., St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Oklahoma Heart, Oklahoma City, Oklahoma
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Providence Cardiology LLC, Columbia, South Carolina
  - Baptist Memorial Hospital, Memphis, Tennessee
  - VA North Texas Health Care System, Dallas, Texas
  - CHI St. Luke's Health / Baylor St. Luke's Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - U of TX Health Science Center San Antonio (UTHSCSA), San Antonio, Texas
  - Trinity Mother Frances/Cardiovascular Associates of East Texas PA, Tyler, Texas
  - Sentara Cardiovascular Research Institute / Norfolk General, Norfolk, Virginia
- Heart Center Alfred Hospital, Melbourne, Victoria, Australia
- Auckland City Hospital, Auckland, New Zealand

REFERENCES:
- [Derived] Mehran R, Faggioni M, Chandrasekhar J, Angiolillo DJ, Bertolet B, Jobe RL, Al-Joundi B, Brar S, Dangas G, Batchelor W, Prasad A, Gurm HS, Tumlin J, Stone GW. Effect of a Contrast Modulation System on Contrast Media Use and the Rate of Acute Kidney Injury After Coronary Angiography. JACC Cardiovasc Interv. 2018 Aug 27;11(16):1601-1610. doi: 10.1016/j.jcin.2018.04.007. PMID 30139467

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Treatment: Standard of Care with the AVERT system
  AVERT
Period: Overall Study
Arm/Group | Active Treatment | Standard of Care
Started (Subjects that signed consent and were randomized.) | 292 | 286
Completed Procedure | 283 | 284
Completed | 269 (9 subjects did not proceed onto procedure in this arm.) | 280 (2 subjects did not proceed onto procedure in this arm.)
Not Completed | 23 | 6
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Death | 4 | 2
Not completed — Lost to Follow-up | 7 | 1
Not completed — See clarification above in comments | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Standard of Care | Total
Number analyzed (Participants) | 292 | 286 | 578
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (9.3) | 72.3 (9.4) | 71.6 (9.4)
Gender [Count of Participants; unit: Participants]
  Female | 114 | 113 | 227
  Male | 178 | 173 | 351

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint
Description: Reduction in the incidence of Contrast Induced Nephropathy (CIN) by evaluating Serum Creatinine levels in subjects for up to 5 days.
Time Frame: 3-5 days
Population: Only subjects that completed blood draws were analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Standard of Care
Number analyzed (Participants) | 281 | 282
Participants | 76 | 75

2. Primary Outcome: Primary Safety Endpoint- Number of Participants Experiencing a Device Related Serious Adverse Event
Description: Analyze the incidence of device related serious adverse events within the treatment arm.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Standard of Care
Number analyzed (Participants) | 292 | 0
Participants | 1 |

3. Secondary Outcome: Secondary Endpoint 1-
Description: Comparison in contrast media volume required between active treament and standard of care.
Time Frame: 30 Days
Population: Reduction in volume of contrast was analysed in an interim analysis once half the patient population was enrolled. Additionally, only subjects that completed the procedure were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: Contrast Volume (ml)
Arm/Group | Active Treatment | Standard of Care
Number analyzed (Participants) | 147 | 137
Contrast Volume (ml) | 87 (52.4) | 102.4 (74.1)

4. Secondary Outcome: Secondary Endpoint 2- Comparison of Serious Adverse Events.
Description: Comparing event rates of serious adverse events 30 days following the index procedure.
Time Frame: 30 Days
Measure: Number; unit: events
Arm/Group | Active Treatment | Standard of Care
Number analyzed (Participants) | 292 | 286
events | 43 | 46

5. Secondary Outcome: Secondary Endpoint 3- Change in Kidney Function.
Description: Change in kidney function by analyzing eGFR 3 to 5 days post procedure.
Time Frame: 3-5 days
Measure: Mean (Standard Deviation); unit: mL/min/1.73m²
Arm/Group | Active Treatment | Standard of Care
Number analyzed (Participants) | 281 | 282
mL/min/1.73m² | 6.3 (8.1) | 5.9 (7.5)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Active Treatment | Standard of Care
Serious Adverse Events (participants affected / at risk) | 36/292 | 38/286
Other Adverse Events (participants affected / at risk) | 0/292 | 0/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=292) | Standard of Care (N=286)
Myocardial Infarction (Cardiac disorders) | 4 (4) | 7 (7)
Dialysis dependent CIN (Renal and urinary disorders) | 3 (3) | 1 (1)
Unplanned re-hospitalization (General disorders) | 26 (28) | 23 (23)
Major bleeding (Surgical and medical procedures) | 6 (6) | 4 (5)
Stroke (Cardiac disorders) | 1 (1) | 0 (0)
All-Cause Mortality (General disorders) | 5 (5) | 3 (3)
Revascularization of target lesion (Cardiac disorders) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No